CLINICAL TRIAL: NCT01026116
Title: Comparing EC-wP Versus EP-wP as Adjuvant Therapy for Breast Cancer Patients Less Than 40 Years Old
Brief Title: A Randomized Trial Comparing EC-wPversus EP-wP as Adjuvant Therapy for Operable Breast Cancer Patients Less Than 40 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of Breast Surgery Department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHBCC09007
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EC-wP (Active Comparator): epirubicin/cyclophosphamide followed weekly paclitaxel
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel
- EP-wP (Experimental): epirubicin/paclitaxel followed by weekly paclitaxel
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Epirubicin — 75 mg/m2 every-3-week for four cycles
Drug: Cyclophosphamide — 600 mg/m2 every-3-week for four cycles
Drug: Paclitaxel — 175 mg/m2 every-3-week for four cycles followed by weekly paclitaxel (80 mg/m2) for 12 weeks

SUMMARY:
Manifold data revealed that young breast cancer patients are characterized by aggressive clinical history. The purpose of this study is to evaluate the efficacy and safety of different strategies incorporating paclitaxel to anthracycline-based regimens in young breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age 18~40
* Unilateral, operable, histologically confirmed adenocarcinoma of the breast
* Stage I-III
* Primary surgery with clear margins plus axillary dissection
* Able to start protocol Rx within 8 weeks of surgery
* Histological or cytological confirmation of estrogen-receptor positive (ER+) breast cancer: the immunohistochemical cut-off for ER positive status was

  1% or more staining in nuclei
* HER-2 negative (IHC 0,1+ or 2+ with a negative in situ hybridization test by chemotherapy
* pathologically confirmed regional node-positive disease, or node-negative disease with high-risk factors (primary tumor diameter >10 mm when histological grade III, or tumor diameter >20 mm when histological grade II)
* ECOG performance status 0-1
* Adequate cardiac, renal, hepatic and hematologic function

Exclusion Criteria:

* Metastatic disease
* Bilateral breast cancer (synchronous or metachronous)
* Prior radiation therapy, hormonal therapy and chemotherapy for breast cancer
* Previous cancer (except treated basal cell and squamous cell carcinoma of the skin or cancer of the uterine cervix)
* HER-2 positive (IHC 3+ OR FISH+) and or triple-negative breast cancer
* Documented history of cardiac disease contradiction anthracyclines
* Concurrent serious illness
* Peripheral neuropathy of CTC grade>1
* History of hypersensitivity to drugs formulated in Cremophor EL polyoxyethylated castor oil), the vehicle used for commercial paclitaxel formulations
* Pregnancy or lactation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 521 (Actual)
Dates: Start 2009-12; Primary Completion 2016-01 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
disease-free survival | every one year
menstrual resumption rate | 12 months after chemotherapy
  Resumption of menses was defined as at least 2 consecutive menstruations, or at least 1 menstruation with a confirmed premenopausal level of FSH and estradiol after chemotherapy

SECONDARY OUTCOMES:
overall survival | every one year

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Principal Investigator — Cancer Hospital, Fudan University
Locations (1):
- Department of Breast Surgery, Cancer Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Derived] Yu KD, Ge JY, Liu XY, Mo M, He M, Shao ZM; SPECTRUM Investigators. Cyclophosphamide-Free Adjuvant Chemotherapy for Ovarian Protection in Young Women With Breast Cancer: A Randomized Phase 3 Trial. J Natl Cancer Inst. 2021 Oct 1;113(10):1352-1359. doi: 10.1093/jnci/djab065. PMID 33822134